CLINICAL TRIAL: NCT04049214
Title: Feasibility Study to Determine the Effect of Meditation on Perioperative Pain and Distress in Newly Diagnosed Breast Cancer Patients
Brief Title: Perioperative Mindfulness Proposal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 173-18-CA
Record Dates: First submitted 2019-07-31; First posted 2019-08-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; DCIS
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditation (Other): Two guided meditations will be provided to participants. They will be asked to meditate twice daily, once in the morning once before bed, for a total time of 12 minutes per day. Surgical treatment and postoperative care will be provided by surgeon preference and usual practice, including post-operative pain medications. For 12 weeks patients will maintain a daily meditation log, medication log and complete daily pain assessment questionnaire.
  Interventions: Other: Meditation

INTERVENTIONS:
Other: Meditation — Two guided meditations will be provided to participants. They will be asked to meditate twice daily, once in the morning once before bed, for a total time of 12 minutes per day. Surgical treatment and postoperative care will be provided by surgeon preference and usual practice, including post-operative pain medications. For 12 weeks patients will maintain a daily meditation log, medication log and complete daily pain assessment questionnaire.

SUMMARY:
The purpose of this study is to determine if a regular meditation and breath work practice started before surgery and continued through post-surgical recovery can improve anxiety and pain related to breast cancer and its treatment.

DETAILED DESCRIPTION:
Breast cancer affects 1 in 8 women in the United States and the majority are managed surgically as part of their primary treatment. Annually over 800 women at Hoag are treated surgically for breast cancer.

Anxiety and fear are commonly associated with breast cancer diagnosis, with as many as 20% of breast cancer patients suffering from full blown depressive disorder and 10% from an anxiety disorder.(1) Mindfulness practices have demonstrated improvements in self reported well being, reductions in stress and fatigue, reduced reactivity to distressing thoughts and improvements in both sensory and affective pain components in a variety of chronic pain conditions including arthritis and chronic pain syndromes. (2) Adoption of Mindfulness Based Stress Reduction (MBSR) has shown improvements in psychological health for breast cancer survivors, (3) but significant reductions in pain levels have not been demonstrated. The limitations of MBSR (Mindfulness Based Stress Reduction) include significant time investment for patients as well as time and cost of care providers and health care systems. The effect of meditation and specific yogic breath work practices on pain has not been studied.

Opioid addiction is a growing social problem. In 2016 over 2 million Americans over the age of 12 were estimated to suffer from addiction to prescription pain medications, leading to over 20,000 overdose related deaths. (4) The majority of these patients were women. Indicated use narcotic exposure has been reported as an initiation event for some patients in the development of opioid addiction, with over 5% of patients who initiated prescription pain medication at the time of surgery continuing to use the medications after the acute surgical process has resolved. (5) We propose to study the effect of meditation and breath work practice on the distress and perioperative pain of breast cancer patients undergoing primary surgical treatment for breast cancer. The benefit of meditation and breath work practice over standard MBSR practice includes lower burden on patients of time and therefore higher potential cost effectiveness and long term sustainability of patients adopting and committing to a regular practice. The breath work and specific meditation practices that will be taught could be a novel method to address perioperative pain, plus improve management of anxiety and stress during this period and beyond. If successful, this pre recorded meditation guidance that patients can utilize in home practice could be a cost effective addition to improve overall perioperative patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age or older
* Subject must be able to speak and read English
* Newly diagnosed with primary breast cancer
* Will receive primary surgical treatment for their breast cancer diagnosis.
* Undergoing lumpectomy with or without autologous reconstruction with or without contralateral surgery for symmetry with or without IORT or simple mastectomy without reconstruction
* Breast cancer or DCIS

Exclusion Criteria:

* Recurrent breast cancer
* Current or history of major psychiatric diagnosis.
* Subjects who are receiving neo-adjuvant chemotherapy
* Subjects undergoing modified radical mastectomy or reconstruction
* Subjects regular meditation practice within the past 12 months (defined as greater than twice weekly practice)
* Subjects unwilling or unable to complete study materials or comply with study visits
* Subjects with no access to email or a mobile phone (required to access meditations)
* Subjects undergoing surgery outside Hoag
* Subjects who have narcotic dependence as defined by regular weekly narcotic use before cancer diagnosis.
* Re-excision after lumpectomy (subjects who require re-excision after initial enrollment will be excluded from final analysis and dropped from the study).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1. Females 18 years of age or older
Enrollment: 24 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Will daily meditation change pain in undergoing primary surgical treatment for newly diagnosed breast cancer, utilizing the MD Anderson Cancer Center Brief Pain Inventory (short form) | 12 weeks
  Baseline pain assessment will be administered after informed consent is obtained. One week before definitive breast cancer surgery research subjects will complete a one on one education session regarding meditation practice with a wellness coach (AW), and complete a baseline NCCN distress survey. They will begin a daily meditation practice.
  Two guided meditations will be provided to participants. They will be asked to meditate twice daily, once in the morning once before bed, for a total time of 12 minutes per day. Surgical treatment and postoperative care will be provided by surgeon preference and usual practice, including post-operative pain medications. For 12 weeks patients will maintain a daily meditation log, medication log and complete daily pain assessment questionnaire using the MD Anderson Cancer Center Brief Pain Inventory (short form)

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States